CLINICAL TRIAL: NCT03567421
Title: Ureteral Stenting After Ureteroscopy for Stone Treatment, A Global Perspective on Indications and Outcomes
Status: Completed | Type: Observational
Sponsor: Société Internationale d'Urologie (Other)
Responsible Party: Sponsor
Other Study IDs: uCARE 2018-001
Record Dates: First submitted 2018-04-26; First posted 2018-06-25 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Stone;Renal; Stone, Kidney; Stone Ureter
Keywords: stone disease; ureteral stent; stenting; ureteroscopy treatment; stent placement; postoperative ureteral stenting; Société Internationale d'Urologie; uCARE
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Ureterolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The exit strategy after ureteroscopy for stone treatment remains a topic for discussion. Current EAU guidelines on urolithiasis state that postoperative stenting is indicated in patients at increased risk of postoperative complications. Stenting is not considered necessary in all other cases, and after uncomplicated procedures.

Objective: To analyse the postoperative ureteral stenting strategy in clinical practice looking at the indication, type of stents used and the duration of stenting after ureteroscopy for stone treatment. Furthermore, the investigators will examine in what setting the stents are being removed postoperatively.

Study design: This study is a prospective, observational, international, multicentre registry study executed by uCARE.

Study population: All patients >18 years with a ureter or renal stone who are planned for ureteroscopic treatment by semi-rigid and/or flexible ureteroscopy are eligible for this study.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The majority of patients with stones receive an indication for its active removal by ureteroscopy. In the last two decades, endourological treatment techniques have evolved with several technological advances through miniaturisation of ureteroscopes, digital improvements, and optical imaging enhancement techniques leading to a better image quality, and the development of different disposables such as single-use digital ureteroscopes. This advancement has led to an increased number of indications for ureteroscopic treatment. Aside from this, there are no specific contraindications for ureteroscopic treatment, apart from general problems such as being unfit for anaesthesia or the presence of urinary tract infections, according to the EAU guidelines.

The indications for active stone removal of ureteral stones include persistent pain or obstruction, renal insufficiency, and in cases when spontaneous passage is less likely. The indications for active removal of renal stones include stone growth, stone formation in patients who are at high risk for stone formation, symptomatic patients, infection, obstruction, stones larger than 15 mm and the comorbidity profile, social situation and preference of the patient.

The procedure can be performed using semi-rigid instruments, mainly for ureter stones, and/or by flexible ureteroscopes, for complete inspection and treatment of the upper tract.

The exit strategy after stone treatment varies depending on patient characteristics and comorbidity, residual stone load, per-operative details and complications, and surgeons' preference. Stent placement is recommended by the EAU guidelines in case of increased postoperative complications; in cases of residual fragments, bleeding, perforation, pregnancy or urinary tract infections; as well as in all doubtful cases to avoid stressful emergencies.

Postoperative stenting increases postoperative morbidity and urologists should carefully balance the pros and cons of postoperative stenting in each individual case. The ideal stent duration is not known. Ureteral stents are usually removed 1-day postoperatively and most urologists will remove double Js 1-2 weeks postoperatively.

It remains a matter of debate whether to stent a patient postoperatively after a ureteroscopic procedure despite the EAU guidelines statement that routine stenting after an uncomplicated procedure with complete stone removal is not necessary.

STUDY OBJECTIVES

The aim of this registry is to review current clinical practice on postoperative ureteral stenting after ureteroscopy for stone treatment. The investigators will explore the answers to the following questions: What are the indications, predictors and outcomes for stent placement? What types of stents are used and what is the duration for stent placement? Hence, the investigators will assess in what setting the stents are being removed, looking at instrumentation, anaesthetics, and location.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old
* Patient is a candidate for ureteroscopic treatment of a ureter or renal stone by semi-rigid and/or flexible ureteroscopy

Exclusion Criteria:

* Patient <18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients >18 years old with a ureter or renal stone that are planned for ureteroscopic treatment are eligible for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 2348 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of patients receiving an internal drain following treatment for urinary stones by ureteroscopy | 6 months
  This number will be reported as a % of the total patients enrolled.

SECONDARY OUTCOMES:
Number of patients requiring secondary interventions [N] | 6 months
  Post-operative secondary interventions include JJ placement, ureter splint placement, nephrostomy tube placement, reURS, clot removal, pharmacological intervention, or other.
Number of patients requiring pain medication at discharge [N] | 6 months
  Pain defined as that requiring additional therapy or pain medication, or prolonged hospital stay due to pain.
Duration of the actual internal drain indwelling time [days] | 6 months
  This number is auto-calculated based from the date of surgery, and date of stent removal or post-operative visit (if no stent was used)
Duration of the internal drain indwelling time as indicated by the surgeon [days] | 6 months
  Calculated as number of days.
% of patients who required anaesthesia for stent removal [Yes/No] | 6 months
  This intraoperative information will be provided by surgeon to indicate whether anesthesia was required during stent removal. Data to be reported as % of total patients.
Incidence of use of flexible instruments for stent removal following ureteroscopy. | 6 months
  As indicated by treating surgeon [Yes/No response].

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Baard, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Mihir Desai, MD, Study Chair — University of Southern California, United States; Jean de la Rosette, MD, Study Director — Istanbul Medipol University, Istanbul, Turkey
Locations (50):
- University of Minnesota, Minneapolis, Minnesota, United States
- China (6):
  - Guangdong Second Provincial General Hospital, The Third Clinical Medical College of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University and Guangdong Key Laboratory of Urology, Guangzhou
  - Ningbo First Hospital, The Affiliated Hospital of Ningbo University, Ningbo
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Shanghai Changhai Hospital, Second Military Medical University, Shanghai
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
- Greece (5):
  - Aretaieion Hospital, Athens
  - Sismanoglio General Hospital, Athens
  - University of Crete, Department of Urology, Heraklion
  - Department of Urology, University Hospital of Larissa, Larissa
  - 1st Department of Urology, Aristotle University, Thessaloniki
- India (2):
  - Jawahar Lal Nehru (JLN) Medical College, Ajmer, Rajasthan
  - Kulkarni Reconstructive Urology Center, Pune
- Indonesia (6):
  - Department of Urology, Hasan Sadikin Hospital/Padjadjaran University, Bandung
  - Department of Urology, Sanglah Hospital/Udayana University, Denpasar
  - Department of Urology, Cipto Mangunkusumo Hospital/University of Indonesia, Jakarta
  - Department of Urology, Saiful Anwar Hospital/Brawijaya University, Malang
  - Department of Urology, Dr. Soetomo Hospital/Airlangga University, Surabaya
  - Department of Urology, Sardjito Hospital/Gadjah Mada University, Yogyakarta
- Shahid Beheshti Hospital, Hamadan University of Medical Sciences, Hamadan, Iran
- University of Basra, College of Medicine, Urology Department, Basra, Iraq
- Pandya Memorial Hospital, Mombasa, Kenya
- Malaysia (5):
  - Selayang Hospital, Batu Caves
  - Serdang Hospital, Kajang
  - Kuala Lumpur Hospital, Kuala Lumpur
  - University of Malaya, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Department of Urology, St. John Clinical Hospital of Emergency, Bucharest, Romania
- Saudi Arabia (3):
  - International Medical Center, Jeddah
  - King Abdulaziz University, Jeddah
  - Prince Sultan Military Medical City, Riyadh
- Sefako Makgatho Health Sciences University, Ga-Rankuwa, South Africa
- SMG-SNU Boramae Medical Center, Seoul, South Korea
- Taiwan (4):
  - Division of Urology, Department of Surgery, Kaohsiung Veterans General Hospital, Kaohsiung, Kaohsiung City
  - Department of Urology, Cardinal Tien Hospital, New Taipei City
  - Department of Urology, En Chu Kong Hospital, New Taipei City
  - Department of Urology, National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (12):
  - Department of Urology, Cukurova University, Adana, Adana
  - Baskent University, Faculty of Medicine, Department of Urology, Ankara
  - Department of Urology, Gazi University, Ankara
  - Department of Urology, Hacettepe University, Ankara
  - Cerrahpasa School of Medicine Istanbul University, Istanbul
  - Department of Urology, University of Health Sciences, Bağcılar Hospital, Istanbul
  - Istanbul Medipol University, Department of Urology, Istanbul
  - Department of Urology, 9 Eylul University, Izmir
  - Konya Meram Education & Research Hospital, Konya
  - Necmettin Erbakan University, Meram Medical School, Konya
  - Selcuk University Selcuklu Medical School, Konya
  - Department of Urology, Bulent Ecevit University, Zonguldak

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Türk C, Knoll T, Petrik A, et al. EAU Guidelines on Urolithiasis 2016. Available at: https://uroweb.org/wp-content/uploads/EAU-Guidelines-Urolithiasis-2016-1.pdf
- [Background] Legemate JD, Wijnstok NJ, Matsuda T, Strijbos W, Erdogru T, Roth B, Kinoshita H, Palacios-Ramos J, Scarpa RM, de la Rosette JJ. Characteristics and outcomes of ureteroscopic treatment in 2650 patients with impacted ureteral stones. World J Urol. 2017 Oct;35(10):1497-1506. doi: 10.1007/s00345-017-2028-2. Epub 2017 Mar 20. PMID 28321499
- [Background] ICH Harmonised Tripartite Guideline. Guideline for Good Clinical Practice E6(R2). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html. Accessed March 25, 2018.